CLINICAL TRIAL: NCT02773498
Title: Comparison of Medical Results of Testicular Sperm Extraction by Conventional Surgery and Microsurgical Track
Acronym: Microsperm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: procedure is too demanding
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/15/7840
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Azoospermia
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional TESE (Active Comparator): Conventional multiple TESE is performed under general or locoregional anesthesia. Through a small vertical incision in the median scrotal raphe, the skin, dartos muscle, and tunica vaginalis are opened to expose the tunica albuginea. The tunica albuginea is ordinarily incised for about 4 mm at the medium region of the testis. A similar biopsy will be systematically performed in the contralateral testis. The biopsy is analyzed by the biologist in the theatre in order to precise if sufficient spermatozoa is retrieved.
  Interventions: Procedure: conventional TESE
- micro TESE (Experimental): Microdissection TESE is also performed under general or locoregional anesthesia. After the tunica albuginea is opened widely along the antiepididymal border, direct examination of the testicular parenchyma is performed under the operating microscope. An attempt is made to identify individual seminiferous tubules that are larger, more opaque and whiter than other tubules in the testicular parenchyma, which are considered to contain spermatozoa. The extracted tubules are analyzed by the biologist in the theatre. The procedure is terminated when sperm are retrieved or further biopsy is thought likely to jeopardize the blood supply of the testis. If all tubules are seen to have an identical morphological appearance, at least three samples (upper, middle, and lower) are obtained. A similar microTESE will be systematically performed in the contralateral testis
  Interventions: Procedure: Micro TESE

INTERVENTIONS:
Procedure: conventional TESE — usual procedure for sperm extraction
  Other Names: conventional surgery
  Arms: conventional TESE
Procedure: Micro TESE — procedure of extraction is performed under the operating microscope
  Other Names: Microdissection surgery
  Arms: micro TESE

SUMMARY:
To compare mobile sperm extraction rate between microTESE and conventional TESE in 18-50 years-old men with non obstructive azoospermia.

DETAILED DESCRIPTION:
About one in ten couples cannot have children without medical assistance. Male factors for infertility are identified in half cases with 10% azoospermia, non-obstructive in most cases. Up to date, testis surgical sperm retrieval for use in ICSI-IVF is the only possibility for those men to have children with their own sperm. Several options are available for surgically retrieving sperm from testis: During conventional testicular sperm extraction (cTESE), the testis is exposed through a small incision, then 1 or more biopsies are randomly made. Up to date, cTESE is considered as the gold-standard for sperm extraction in this population.

However, the success of surgical sperm extraction concerns a man out of two having cTESE for non-obstructive azoospermia.

On the other hand, Schlegel showed in 1997 that cTESE induces a significative loss of testicular tissue with possible impact on male endocrine balance with occurence of hematomas, inflammatory reshuffles and ischaemic lesions, compromising some regions in the testicular parenchyme. Another option for surgical sperm extraction is micro-surgery called microTESE (or µTESE). It consists in examining the testicular parenchyme under a high-power microscope (up to 25 magnification), screening for white opaque tubules with higher diameter which indicates possible active spermatogenesis. The benefits of µTESE are: (1) a better identification of sites of sperm production in the testis, (2) a better preservation of testicular vasculature decreasing the risk of postoperative hematoma or tissue ischemia and (3) excision of 3 to 10 times less tissue.

Nevertheless, no randomized studies have compared both techniques to validate such an assumption. In 2014, the results of a meta-analysis performed by Deruyver showed that, among the 7 original articles comparing cTESE to µTESE, 3 were retrospective studies and the remaining 4 prospective studies were not randomized.

It is highly unlikely that this better outcome is related to patient selection. Nevertheless, the relatively small number of studies comparing both methods makes it difficult to draw definitive conclusions This study is based on the hypothesis that µTESE is a superior technique than cTESE with a difference of 20% like observed in Deruyver's meta-analysis.

The principal objective is to compare motile sperm extraction rate between μTESE and cTESE in 18-50 years-old men with NOA.

ELIGIBILITY:
Inclusion Criteria:

* 2 consecutive spermograms (with ±3 months interval) confirming absence of sperm (azoospermia)
* diagnosis of non-obstructive azoospermia on the basis of a complete history, physical examination, endocrine profile, ultrasound and chromosomal analysis

Exclusion Criteria:

* History of previous testicular surgery, except orchiopexy for undescended testis.
* Monochordy
* Ultrasound revealed testicular nodule
* Y chromosome microdeletions type AZFa and b.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
sperm extraction | time of surgery
  positivity (presence, coded 1) or negativity (absence, coded 0) of the sperm extraction, based on possibility of having at least 1 mobile sperm

CONTACTS AND LOCATIONS:
Overall Officials: Eric Huyghe, MD, PhD, Principal Investigator — U H Toulouse
Locations (5):
- France (5):
  - University Hospital, Bordeaux
  - University Hospital, Lille
  - University Hospital, Paris
  - University Hospital, Rouen
  - University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsujimura A, Matsumiya K, Miyagawa Y, Tohda A, Miura H, Nishimura K, Koga M, Takeyama M, Fujioka H, Okuyama A. Conventional multiple or microdissection testicular sperm extraction: a comparative study. Hum Reprod. 2002 Nov;17(11):2924-9. doi: 10.1093/humrep/17.11.2924. PMID 12407050